CLINICAL TRIAL: NCT02698670
Title: Prospective Registry on User Experience With The Mapping System For Ablation Procedures
Acronym: TRUE-HD
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 91118280
Record Dates: First submitted 2016-02-24; First posted 2016-03-04 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2017-06

CONDITIONS: Cardiac Arrhythmias
Keywords: Cardiac Arrhythmias; Cardiovascular Disease; Radiofrequency Ablation; Cardiac Mapping
MeSH Terms: conditions — Arrhythmias, Cardiac; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Rhythmia mapping system — A 3-D Cardiac Mapping system
Device: IntellaMap Orion mapping catheter — A diagnostic basket mapping catheter

SUMMARY:
This is an observational, prospective, non-randomized, multicenter, post approval study being conducted in the United States, Europe and Asia-Pacific Regions.

DETAILED DESCRIPTION:
The TRUE HD Study is aimed at collecting real-world data on the use of the Rhythmia mapping system and the IntellaMap Orion mapping catheter in patients indicated for ablation procedure with use of a 3D Mapping system.

The study will collect specific information on management of ablation procedures with the commercial system including but not limited to acute procedural success, type and proportion of arrhythmias mapped/treated, and how mapping system is used overall. Usage data may be used for the planning of future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are eligible for an ablation procedure with the Rhythmia 3D mapping system and IntellaMap Orion mapping catheter according to current international and local guidelines (and future revisions) and per physician discretion;
* Subjects who are willing and capable of providing informed consent;
* Subjects who are willing and capable of participating in all testing associated with this clinical investigation at an approved clinical investigational center;
* Subjects whose age is 20 years or above, or of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

* Subjects requiring de novo ablation of atrial fibrillation;
* Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments; each instance must be brought to the attention of the sponsor to determine eligibility*;
* The subject is unable or not willing to complete follow-up visits and examination for the duration of the study;
* Subjects who have undergone a previous cardiac ablation within 30 days prior to enrollment;
* Unrecovered/unresolved Adverse Events from any previous invasive procedure;
* Women of childbearing potential who are, or plan to become, pregnant during the time of the study (method of assessment upon physician's discretion).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are eligible for an ablation procedure with the Rhythmia 3D mapping system and IntellaMap Orion mapping catheter according to current international and local guidelines (and future revisions) and per physician discretion
Sampling Method: Probability Sample
Enrollment: 577 (Actual)
Dates: Start 2016-05-25; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Acute Procedural Success | At the end of the index procedure (Day 0)
  Primary endpoint is the acute procedural success for the primary arrhythmia in the whole cohort of ablation procedures. A procedure will be defined successful if all the following conditions will occur during the case: 1) ability to map, 2) completion of the necessary ablation applications, 3) primary arrhythmia termination (when applicable), and 4) validation of ablation through appropriate technique(s).

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Hindricks, Principal Investigator — Gerhard Hindricks
Locations (28):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Hoag Memorial Hospital, Orange, California
  - Torrance Memorial Medical Center, Torrance, California
  - University of Chicago Hospital, Chicago, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - University of Michigan Hospitals, Ann Arbor, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Maimonidies Hospital, New York, New York
  - Strong Memorial Hospital of the University of Rochester, Rochester, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Riverside Methodist - Ohio Health, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Heart Rhythm Institute, Oklahoma City, Oklahoma
  - Oregon Health Sciences University, Portland, Oregon
  - Baptist Memorial Hosptial, Memphis, Tennessee
  - Trinity Mother Francis, Tyler, Texas
  - Virginia Mason Medical Center, Seattle, Washington
- Wesley Medical Research, Brisbane, Queensland, Australia
- France (2):
  - CHU de Bordeaux, Pessac
  - Centre Hôpital Universitaire Rangueil, Toulouse
- Germany (2):
  - Universitaetsklinik Eppendorf, Hamburg
  - Herzzentrum Universität Leipzig, Leipzig
- Queen Mary Hospital, Hong Kong, Hong Kong
- University Medical Center Groningen, Groningen, Netherlands
- Clinica Universitaria de Navarra, Pamplona, Spain
- United Kingdom (2):
  - Harefield Hospital, London
  - The Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: No